CLINICAL TRIAL: NCT02788006
Title: Phase II Study Evaluating the Efficacy and the Safety of Regorafenib in Patients Aged More Than 70 Years Old With a Metastatic Colorectal Adenocarcinoma .
Brief Title: Efficacy and the Safety of Regorafenib in Patients Aged More Than 70 Years With a Metastatic Colorectal Adenocarcinoma .
Acronym: REGOLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FFCD 1404 - REGOLD
Record Dates: First submitted 2016-05-20; First posted 2016-06-02 (Estimated); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Adenocarcinoma
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib 160 mg (Experimental)
  Interventions: Drug: Regorafenib 160 mg

INTERVENTIONS:
Drug: Regorafenib 160 mg

SUMMARY:
Multicenter prospective phase II study evaluating regorafenib in older patients with metastatic colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer with histological proof
* Measurable disease according RECIST 1.1
* Age ≥ 70 years
* ECOG ≤ 1
* Biological values Haemoglobin ≥ 9 g/dL, PNN ≥ 1500/mm3, platelets≥ 100 000/mm3, bilirubin ≤ 1,5N, ASAT, ALAT et PAL ≤ 2,5N (≤ 5N if hepatic metastases), lipase ≤1,5N, TP≥ 70%, Creatinine clairance ≥ 30 mL/min
* Patient without response to 5FU chemotherapy or anti-vegf treatment or anti EGFR treatment (if RAS wild-type), in progression during this treatment or treatment stopped because of toxicities
* Geriatric Questionnaires answered
* Life-expectancy ≥ 3 months
* Informed Consent Signed

Exclusion Criteria:

* Not able to swallow tablets (crushed tablets are not allowed)
* Previous treatment with regorafenib or other multikinase treatment
* Other cancer during the last 5 years, excepted in-situ cervix cancer, skin cancer non melanoma and cancer of the bladder curatively treated
* Radiotherapy: with extended fields in the last 4 weeks, with limited fields in the last 2 weeks previous inclusion
* Toxicity > grade 1 not resolved with previous treatment
* Major surgery in the 28 days before the inclusion
* Non cicatrized injury, ulcer or bone fracture
* Congestive Cardiac insufficiency classe >2 (NYHA)
* Unstable angor in the last 3 months
* Myocardial Infraction in the 6 months before inclusion
* HTA not controlled
* Pheochromocytome
* Arterial or venous thromboembolism in the past 6 months
* Infection of grade > 2
* VIH infection
* B or C hepatitis necessiting a specific treatment
* Cirrhosis
* Suspicion of brain metastasis or brain metastasis
* Haemorraghe ofgrade >3 in the last weeks
* Symptomatic Pulmonary fibrosis
* Proteinuria > grade 3
* Malabsorption
* Allergy know to the treatment or to one similar treatment or to one treatment component
* Systemic anti-cancer drug during the study or the the last 4 weeks
* Concomitant treatment with CYP3A4 inhibitor or inductor or with UGT1A9 inhibitor
* Social, psychological or medical condition which can interfere with the study participation

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas APARICIO, Pr, Principal Investigator — Hôpital Avicenne BOBIGNY
Locations (16):
- France (16):
  - CH Victor Dupouy, Argenteuil
  - Centre François Bacless, Caen
  - Centre Oncologie et Radiothérapie, Dijon
  - Clinique du Cap d'Or, La Seyne-sur-Mer
  - Caluire et Cuire - Infirmerie Protestante de Lyon, Lyon
  - CH Lyon Sud (HCL) - Pierre Benite, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Hôpital Européen, Marseille
  - CHRU - Hôpital Saint Eloi, Montpellier
  - CHR - Service HGE, Orléans
  - Saint Joseph, Paris
  - CH, Perpignan
  - Hôpital Haut Leveque, Pessac
  - CH Annecy Genevois, Pringy
  - Centre Paul Strauss, Strasbourg
  - Hôpital privé, Villeneuve-d'Ascq

REFERENCES:
- [Result] Aparicio T, Darut-Jouve A, Khemissa Akouz F, Monterymard C, Artru P, Cany L, Romano O, Valenza B, Le Foll C, Delbaldo C, Falandry C, Norguet Monnereau E, Ben Abdelghani M, Smith D, Rinaldi Y, Pere Verge D, Baize N, Maillard E, Dohan A, Des Guetz G, Pamoukdjian F, Lepage C. Single-arm phase II trial to evaluate efficacy and tolerance of regorafenib monotherapy in patients over 70 with previously treated metastatic colorectal adenocarcinoma FFCD 1404 - REGOLD. J Geriatr Oncol. 2020 Nov;11(8):1255-1262. doi: 10.1016/j.jgo.2020.04.001. Epub 2020 Apr 22. PMID 32334940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2016 to April 2017, 43 patients were enrolled in the trial by 25 centers in France.
Pre-assignment Details: Before enrollement, standard examinations (biological, clinical, ECG) as well as geriatric questionnaires were done. In terms of imaging, abdominal and thoracic computed tomography scan or MRI were also done.
Groups:
- Regorafenib 160 mg: Regorafenib monotherapy at an initial dose of 160 mg once daily orally (21 days on, 7 days off treatment)
Period: Overall Study
Arm/Group | Regorafenib 160 mg
Started | 43
Completed | 42
Not Completed | 1
Not completed — Patient not treated | 1

BASELINE CHARACTERISTICS:
Population: All the patients enrolled in the study and treated by Regorafenib
Arm/Group | Regorafenib 160 mg
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.9 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 42
Region of Enrollment [Number; unit: participants]
  France | 42
Koehne Score [Count of Participants; unit: Participants] — Low is for patients with OMS equal to 0 or 1 and with 1 metastatic site
  Intermediate is for patients with 0MS equal to 0-1 and with more than 1 metastatic site and Phosphatases Alcalines <300 U/L, or patients with OMS >1 and WBC <10.109/L and 1 metastatic site
  Higi is for patients with OMS 0/1 and with more than 1 metastatic site and with phosphatases alcalines > 300 U/L or patients with OMS > 1 and with more than 1 metastatic site or patients with WBC >10.109 /L
  Participants
    Low | 16
    Intermediate | 22
    High | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Tumoral Control Rate at 2 Months
Description: Tumor control rate is defined as the percentage of patients with complete tumor response, partial tumor response, or tumor stability on regorafenib therapy at 2 months after initiation of therapy as determined by the investigator per Response Evaluation Criteria In Solid Tumors Criteria (RECIST V1.1 criteria) for target lesions and assessed by CT-Scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stability : neither complete or partial response nor progression.
Time Frame: 2 months after the start of treatment
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Groups:
- Regorafenib 160 mg: Regorafenib 160 mg
Arm/Group | Regorafenib 160 mg
Number analyzed (Participants) | 35
Percentage of patients | 31.4 [18.7 to 46.6]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of the patient's inclusion to the patient's death (all causes). For alive patients the date of the latest news wastaken into account.
  Overall survival was estimated also after the treatment stopped explaining the difference of time frame between this outcome and the adverse events outcome.
Time Frame: Up to approximatively 1 year after the end of the treatment
Population: All patients included in the study and who have been treated with regorafenib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Regorafenib 160 mg
Number analyzed (Participants) | 42
months | 7.5 [5.5 to 10.6]

ADVERSE EVENTS:
Time Frame: Up to the end of treatment. Treatement was usually stopped after 70 days of treatments. Overall survival was estimated also after the treatment stopped explaining the difference of time frame between this outcome and the adverse events outcome.
Arm/Group | Regorafenib 160 mg
All-Cause Mortality (participants affected / at risk) | 36/42
Serious Adverse Events (participants affected / at risk) | 17/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib 160 mg (N=42)
Pulmonary embolism (Vascular disorders) | 1
Fall (Injury, poisoning and procedural complications) | 3
Hypertension (Cardiac disorders) | 2
Haematoma (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Cerebrovascular ischemia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Fatigue (General disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 1
Deshydratation (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regorafenib 160 mg (N=42)
Aspartate aminotransferase increased (Investigations) | 21
Alanine aminotransferase increased (Investigations) | 12
Total Bilirubin increased (Investigations) | 22
Gamma-glutamyltransferase increased (Investigations) | 31
White blood cell count decreased (Investigations) | 4
Lipase increased (Investigations) | 7
Neutrophils decreased (Investigations) | 4
Lymphocytes decreased (Investigations) | 3
Phosphatases Alcalines increased (Investigations) | 21
Platelets decreased (Investigations) | 20
Hypertension (Cardiac disorders) | 12
Anemia (Blood and lymphatic system disorders) | 19
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11
Headache (Nervous system disorders) | 3
Dysgueusia (Nervous system disorders) | 4
Fatigue (General disorders) | 34
Pyrexia (General disorders) | 7
Constipation (Gastrointestinal disorders) | 13
Diarrhoea subjects (Gastrointestinal disorders) | 17
Abdominal pain (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 5
Proteinuria (Renal and urinary disorders) | 9
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Hypokaliemia (Metabolism and nutrition disorders) | 3
Hypothyroidism (Endocrine disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 23
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Musculoskeletal and connective tissue disorders) | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT02788006/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT02788006/SAP_001.pdf